CLINICAL TRIAL: NCT06768372
Title: Investigation of the Relationship Between Temporomandibular Joint Dysfunction Prevalence and Oral Habits, Food Consumption Frequency and Eating Behaviour in University Students: A Cross-Sectional Study
Brief Title: Temporomandibular Joint Dysfunction Prevalence and Oral Habits, Food Consumption Frequency and Eating Behaviour
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Principal Investigator, Karadeniz Technical University
Other Study IDs: KTU-FTR-2024/150
Record Dates: First submitted 2024-12-24; First posted 2025-01-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Joint Disorders; Oral Habits; University Students
Keywords: Temporomandibular Joint Dysfunction; Oral Habits; Food Consumption; Eating Behaviour
MeSH Terms: conditions — Temporomandibular Joint Disorders; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: University students

SUMMARY:
This study was planned to investigate the prevalence of TMD in university students and to determine possible predisposition factors by evaluating oral habits, food consumption frequency and eating behaviors thought to be related to TMD.

DETAILED DESCRIPTION:
No study has been found examining the relationship between temporomandibular joint dysfunction (TMD) and oral habits, food consumption frequency and eating behavior. In this context, it is thought that understanding the relationships mentioned may provide different perspectives and help develop an effective treatment program.

ELIGIBILITY:
Inclusion Criteria:

1. Continuing undergraduate education at faculties/colleges affiliated with Karadeniz Technical University
2. Being able to read and write in Turkish
3. Agreeing to participate in the study

Exclusion Criteria:

1. Having a local or systemic disease that may affect oral and jaw health
2. Having had an operation / trauma to the cervical region or TMJ

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Presence and Severity of Temporomandibular Dysfunction | an average of 6 months
  Fonseca Anamnestic Index, reported as a reliable and valid index, will be used to determine the presence and severity of TMD. The total score ranges from 0 to 100. The total score of the index allows the following classification: no TMD (≤ 15), mild TMD (20-40), moderate TMD (45-65), and severe TMD (70-100).

SECONDARY OUTCOMES:
Oral Habits | an average of 6 months
  The Oral habits checklist, a questionnaire recommended for the assessment of parafunctional behaviors, will be used.
Food Consumption Frequency | an average of 6 months
  The frequency and amount of food groups or nutrients consumed will be questioned. Frequency of consumption can be given as day, month or week.
Eating Behavior | an average of 6 months
  The Adult Eating Behavior Scale will be used. There are 8 sub-dimensions and a total of 35 items in the scale. It is scored with a five-point Likert. The score obtained shows the tendency towards the relevant behavior. There is no scale measuring the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical Univerity, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No